CLINICAL TRIAL: NCT02914197
Title: Giving Information on the Risks and Limitations of Mammography Screening (GIRLS): a Randomized Controlled Trial
Brief Title: Giving Information on the Risks and Limitations of Mammography Screening (GIRLS)
Acronym: GIRLS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McMaster University (Other)
Collaborators: David Braley and Nancy Gordon Chair in Family Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 2016-001
Record Dates: First submitted 2016-09-22; First posted 2016-09-26 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2017-08

CONDITIONS: Breast Neoplasm
Keywords: Decision; Mammography; Informed Choice; Full Information; Decision Aid; Self-efficacy; Shared decision making; Over-detection; Over-diagnosis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Full information (Experimental): The intervention arm will receive full information on the risks and benefits of mammography through:
  1. Decision aid
  2. YouTube video
  3. Group information session
  Interventions: Other: Full information
- Control (No Intervention): Standard information leaflet for breast screening from Cancer Care Ontario

INTERVENTIONS:
Other: Full information — Patients will be randomized to receive full information or standard information at the study start. The second wave will follow the same randomization process 6 months following the study start.
  Arms: Full information

SUMMARY:
To trial the provision of full information on the benefits and risks of mammography in women that are eligible for breast screening. The knowledge many women have of mammography is not reflective of the recent change in evidence; it is often missing information on over-diagnosis and over-detection. Women tend to overestimate their risk of breast cancer and the benefits of breast screening. In addition, universal breast screening programs are biased towards emphasizing screening. However, a mammogram is not a perfect test and there is no right or wrong decision about whether to have a screening mammogram. It is an individual woman's decision to make. To understand the effect of changing information to reflect the potential for over-diagnosis and over-treatment, we will carry out a pragmatic controlled trial of implementation of balanced information on mammography in family practice.

DETAILED DESCRIPTION:
1:1 double-blinded randomized controlled trial of patients to receive the intervention or standard information (control) at the study start in an information package. The intervention includes a decision aid (previously developed by Hersch et al. 2015, with minor modifications to reflect the Canadian context), a YouTube video link and an invitation to attend a group information session. The intervention or standard information, depending on participants assigned study group, will be mailed or emailed to participants. The information packages will also include questionnaires to collect data on outcome measures. There will be two study waves to account for women's eligibility at different time points (i.e. when approaching a mammogram due date). The first wave of participants will receive their information package at the study start and the second wave of participants will be sent their information packages 6 months after the study start. Each wave of participants will be followed for one year. Data collection will include quantitative measures of factors relevant to the decision-making process. Screening participant rates will be measured for each wave of participants, 6 months and 12 months after their respective enrollment date. Qualitative methods will be used to obtain an understanding of clinician's perception of decision aids in a primary care setting. Outcome measures and analyses will be blinded.

ELIGIBILITY:
Inclusion Criteria:

* Patient on the active roster of physicians of MUSIC (McMaster University Sentinel and Information Collaboration; McMaster Family Health Team).
* Due for a mammogram (have not had a mammogram ≥ 18 months) according to Canadian screening interval recommendations for routine screening.

Exclusion Criteria:

* Previous history of invasive or non-invasive breast cancer.
* At higher risk for breast cancer compared to the general population i.e. identified as having the BRCA1 or BRCA2 gene, immediate family member has had breast cancer.
* Have had a mammogram within the last 18 months (< 18 months).

Ages: 47 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 608 (Estimated)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Self-efficacy | 1 month
  Decision Self-Efficacy Scale

SECONDARY OUTCOMES:
Informed Choice (Knowledge) | 1 month
  Informed choice is comprised of knowledge, attitudes and intention/decisions. Informed choice will be measured using intention to screen at the first data collection point and screening participation at the second and third data collection point.
  Knowledge will be measured using the Multidimensional Measure of Informed Choice (MMIC).
Informed Choice (Attitude) | 1 month
  Informed choice is comprised of knowledge, attitudes and intention/decisions. Informed choice will be measured using intention to screen at the first data collection point and screening participation at the second and third data collection point.
  Attitudes will be measured using the Multidimensional Measure of Informed Choice (MMIC).
Informed Choice (Intention) | 1 month
  Informed choice is comprised of knowledge, attitudes and intention/decisions. Informed choice will be measured using intention to screen at the first data collection point and screening participation at the second and third data collection point.
  Intention to screen will be measured using a 5-point Likert scale.
Decisional Conflict | 1 month
  SURE (Decisional Conflict Scale- SURE Test for clinical practice)
Anxiety | 1 month
  Women will be asked about their anxiety towards participating in breast screening after reading their information pamphlet using a 4-point Likert scale.
Trust in Medical System | 1 month
  MMI (Medical Mistrust Index)
Perception of Health Provider Recommendation | 1 month
  Women will be asked to assess their perception of the strength of the recommendation that their health care provider makes with respect to breast screening.
Information Relevant to the Decision Making Process | 1 month
  Women will be asked to describe the information that was relevant to their individual decision making process.
Decision Regret | 12 month
  Decision Regret Scale
Screening Participation | 6 months and 12 months
  Data on a women's decision to undergo screening through mammography will be obtained from patient's electronic medical record.
Acceptance of a Decision Aid in Primary Care | 12 months
  Clinician staff will be asked to list the five best things and five worst things about the implementation of a patient focused decision aid.
Knowledge of the Benefits and Risks of Mammography | 1 month
  Multiple choice question on knowledge of breast cancer mortality reduction and over-diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Department of Family Medicine, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No